CLINICAL TRIAL: NCT06417190
Title: IIT2023-13-BALLAS-VHTMT: Bladder Preservation for Patients With Muscle Invasive Bladder Cancer (MIBC) With Variant Histology
Brief Title: Bladder Preservation for Patients With Muscle Invasive Bladder Cancer (MIBC) With Variant Histology
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leslie Ballas (Other)
Responsible Party: Sponsor-Investigator, Leslie Ballas, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-13-BALLAS-VHTMT
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Tumor
Keywords: Trimodal Therapy (TMT); Neoadjuvant Chemotherapy; muscle-invasive urothelial cell bladder cancer (MIBC)
MeSH Terms: conditions — Neoplasms | interventions — Trail Making Test; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Neoadjuvant chemotherapy followed by trimodal therapy consisting of TURBT followed by concurrent chemotherapy with radiation therapy
  Interventions: Drug: Trimodal therapy (TMT) within 45 days of neoadjuvant chemotherapy (NAC)

INTERVENTIONS:
Drug: Trimodal therapy (TMT) within 45 days of neoadjuvant chemotherapy (NAC) — Single-arm, open-label

SUMMARY:
This is a Phase II, single cohort study designed to evaluate outcomes in patients with muscle invasive bladder cancer (MIBC) with variant histology who receive neoadjuvant chemotherapy (NAC) with or without immunotherapy (IO) followed by trimodal therapy (TMT). Enrolled patients will undergo at least 3 cycles of NAC +/- IO (oncologist's choice) followed by a four- or six-week course of concurrent standard of care chemotherapy and radiation therapy. These patients will be compared with historical controls of patients with a diagnosis of pure urothelial carcinoma who have undergone TMT. This study has been designed to test the hypothesis that variant histology TMT can be delivered within 45 days of NAC +/- IO and is therefore a viable option in patients who are risk of systemic disease spread.

DETAILED DESCRIPTION:
Trimodal therapy (TMT) is accepted as an NCCN category 1 alternative to radical cystectomy (with neoadjuvant chemotherapy) in patients with cT2N0M0 muscle-invasive urothelial cell bladder cancer (MIBC). Not all patients with MIBC have pure urothelial cell carcinoma; urothelial carcinoma with variant histology (VH) described any morphologic variant of conventional urothelial carcinoma that is believed to be derived from urothelial carcinoma and is typically admixed with conventional urothelial carcinoma in the same tumor. Variant histologies described include squamous differentiation, glandular differentiation, micropapillary, sarcomatoid, small cell/neuroendocrine, plasmacytoid and nested variant. This is a rare tumor type and understudied. For patients with variant histologies there is limited data on the use of trimodal therapy. There are a couple single institution retrospective studies and data from the NCDB, but no prospective data.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of MIBC with variant histology, cT2-T4N0M0, confirmed by TURBT and CT C/A/P and/or PET.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Evidence of diffuse cis on pathology
* Presence of bilateral hydronephrosis (if hydronephrosis is present, can only be unilateral)
* Prior radiotherapy to the pelvis
* History of systemic therapy for MIBS
* Presence of concurrent cancer (remote history of cancer (>5 years) allowed if the patient is without evidence of disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of initiating TMT | 45 days
  To evaluate the feasibility of initiating TMT within 45 days of completion of NAC - Feasibility will be defined as at least 17 study participants initiating TMT within 45 days of NAC

SECONDARY OUTCOMES:
3-year bladder intact event free survival (BIEFS) | 3 year
  To estimate 3-year bladder intact event free survival (BIEFS) in patients undergoing TMT for MIBC with VH-TMT

OTHER OUTCOMES:
Progression free (<=T2) survival rates | 3 year
  To estimate progression free (<=T2) survival rates from TMT
Metastasis-free survival | 3 year
  To estimate the metastasis-free survival of TMT
Rate of salvage cystectomy | 3 year
  To estimate the rate of salvage cystectomy following TMT
Blood and urine correlatives of clinical outcomes | 3 year
  To investigate blood and urine correlatives of clinical outcomes (Signatera and Oncuria)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Ballas, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No